CLINICAL TRIAL: NCT05527873
Title: Respiratory Complications of Operated Esophageal Atresia in Children
Acronym: ATRESIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8562
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Esophageal Atresia
Keywords: esophageal atresia; esophageal malformation; gastroesophageal reflux; asthma; bronchial hyperreactivity
MeSH Terms: conditions — Esophageal Atresia; Gastroesophageal Reflux; Asthma; Bronchial Hyperreactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The respiratory complications of esophageal atresia have already been identified.

They are mainly related to tracheomalacia linked to the esophageal malformation, and are aggravated by frequently associated gastroesophageal reflux.

In this context, symptoms of asthma (or bronchial hyperreactivity) occur more frequently than in the general population and persist into adulthood. Their pathogenesis is still poorly understood and is the subject of much discussion.

The therapeutic management of these respiratory complications, poorly codified, remains very heterogeneous from one center to another. In France, the summary of knowledge is updated by the Reference Center for chronic and malformative diseases of the esophagus.

ELIGIBILITY:
Inclusion criteria:

* Child aged 1 to 12 years old
* Child operated on for esophageal atresia between 01/01/2010 and 31/12/2020 and followed up at the University Hospitals of Strasbourg
* Child who has not expressed, after being informed, his opposition to the reuse of his data for the purposes of this research
* Parental authority having not expressed, after being informed, their opposition to the reuse of their child's data for the purposes of this research.

Exclusion criteria:

Subject and/or parental authority having expressed their opposition to participating in the study

Ages: 1 Year to 12 Years | Sex: All
Age Groups: Child
Study Population: Child aged 1 to 12 years old operated on for esophageal atresia and followed up at the University Hospitals of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Retrospective study of respiratory complications of esophageal atresia in children | Files analysed retrospectively from January 01, 2010 to December 31, 2020 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Laurence WEISS, MD, Principal Investigator — Centre de Ressources et de Compétences de la Mucoviscidose (CRCM) - CHU de Strasbourg - France
Locations (1):
- Centre de Ressources et de Compétences de la Mucoviscidose (CRCM) - CHU de Strasbourg - France, Strasbourg, France